CLINICAL TRIAL: NCT02744417
Title: Effect of Smoking Cessation on Clinical and Microbiological Outcomes of the Non-surgical Periodontal Therapy
Acronym: EsCAPE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claudio Mendes Pannuti (Other)
Responsible Party: Sponsor-Investigator, Claudio Mendes Pannuti, Associate Professor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EsCAPE2
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Periodontitis
Keywords: smoking cessation; tobacco; periodontal; subgingival microorganisms
MeSH Terms: conditions — Periodontitis; Smoking Cessation | interventions — Nicotine Replacement Therapy; Nicotine Chewing Gum; Bupropion; Varenicline

STUDY DESIGN:
Masking Description: The outcome assessor was blind to smoking status. Before each follow-up periodontal examination (3, 6 and 12 months), the following procedures were performed by a periodontist: (1) removal of all tobacco stains from subject's teeth and/or dental polishing, with a standardized duration of up to 30 min., (2) 0.12% chlorohexidine rinse (1min.) aimed to hide any possible cigarette odour exhaled from the oral cavity. After these procedures, the examiner entered the examination room fully equipped (including a mask), in order to avoid noticing the smoking status by odour
Oversight: Data Monitoring Committee: No

ARMS (1):
- Smoking cessation therapy (Experimental): Non-surgical periodontal therapy and concurrent smoking cessation therapy, with Smoking cessation counseling, Nicotine replacement therapy, use of bupropion hydrochloride and varenicline
  Interventions: Behavioral: Smoking cessation counseling; Procedure: Non-surgical periodontal therapy; Drug: Nicotine replacement therapy; Drug: bupropion hydrochloride; Drug: Varenicline

INTERVENTIONS:
Behavioral: Smoking cessation counseling — Multidisciplinary smoking cessation counseling, performed by a team comprising physicians, nurses, a psychologist and dentists. It consisted of four 1-h counselling lectures delivered by physicians, psychologist-assisted cognitive behavioural therapy, and counseling provided by dentists during the active phase of the treatment and maintenance session, using motivational interviewing techniques
Procedure: Non-surgical periodontal therapy — Full-mouth supra and subgingival scaling and root planing (with curettes and ultrasonic scaler); oral hygiene instruction and motivation and removal of intra-oral plaque retentive factors
Drug: Nicotine replacement therapy — Nicotine replacement therapy: chewing gum (Nicorette chewing gum 2-4mg) and patches (Nicorette patches 15-25mg)
  Other Names: Nicorette
Drug: bupropion hydrochloride — bupropion hydrochloride 150mg
  Other Names: Zyban
Drug: Varenicline — Varenicline 0,5mg
  Other Names: Champix

SUMMARY:
The aim of this prospective interventional study is to verify the efficacy of smoking cessation on clinical and microbiological outcomes of non-surgical periodontal therapy of chronic periodontitis patients. Smokers willing to quit received periodontal treatment and concurrent smoking cessation therapy. Periodontal maintenance was performed every 3 months. A single calibrated examiner, blinded to smoking status, assessed periodontal clinical outcomes and applied a structured questionnaire in order to collect demographic and behavioural information. Further, expired carbon monoxide concentration were measured with a monoximeter. A pooled subgingival plaque sample was collected from the deepest periodontal pocket from each participant. The presence and quantification of Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia and Treponema denticola were determined using (RT-PCR).

DETAILED DESCRIPTION:
Smokers willing to quit, with 10 teeth or more, and with periodontitis (30% or more of their teeth with proximal attachment loss ≥ 5 mm) were enrolled in the study. All subjects received periodontal treatment and concurrent smoking cessation therapy. Smoking cessation therapy was performed by a team comprising physicians, nurses, a psychologist and dentists, and consisted of four 1-h counselling lectures, psychologist-assisted cognitive behavioral therapy, nicotine replacement therapy and medication (bupropion or varenicline). Smoking cessation motivation was reinforced by dentists at the maintenance sessions, by means of motivational interviewing techniques. Periodontal therapy consisted in full-mouth supra and subgingival scaling and root planing (with curettes and ultrasonic scaler); oral hygiene instruction and motivation and removal of intra-oral plaque retentive factors. Further, periodontal maintenance was performed every 3 months.

A single calibrated examiner, blinded to smoking status, assessed periodontal clinical outcomes (recession, pocket depth, clinical attachment level, plaque index and bleeding on probing). A structured questionnaire was applied in order to collect demographic and behavioral information. Expired carbon monoxide concentration was measured with a monoximeter, in order to validate smoking status. A pooled subgingival plaque sample was collected from the deepest periodontal pocket from each participant. The presence and quantification of Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia and Treponema denticola were determined using real time - PCR (RT-PCR).

ELIGIBILITY:
Inclusion Criteria:

* smokers willing to stop smoking
* >10 teeth
* periodontitis (30% or more of their teeth with proximal attachment loss ≥ 5 mm)

Exclusion Criteria:

* systemic conditions considered as risk factors for periodontal disease,
* periodontal therapy in the last 6 months
* continuous systemic use of anti-inflammatory or steroidal drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-08; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Attachment Level | baseline - 12 months
  Change in Clinical Attachment Level (millimeters) after 12 months

SECONDARY OUTCOMES:
Change in Gingival recession | baseline - 12 months
  Change in Gingival recession (millimeters) after 12 months
Change in Pocket depth | baseline - 12 months
  Change in Pocket depth (millimeters) after 12 months
Change in bleeding on probing | baseline - 12 months
  Change in bleeding on probing (percentage of sites with bleeding) after 12 months
Change in visible plaque | baseline - 12 months
  Change in visible plaque (percentage of sites with visible plaque) after 12 months
Prevalence and levels of Aggregatibacter actinomycetemcomitans | baseline - 12 months
  Prevalence and levels of Aggregatibacter actinomycetemcomitans determined by means of (RT-PCR).
Prevalence and levels of Porphyromonas gingivalis | baseline - 12 months
  Prevalence and levels of Porphyromonas gingivalis, determined by means of (RT-PCR).
Prevalence and levels of Tannerella forsythia | baseline - 12 months
  Prevalence and levels of Tanerella forsythia, determined by means of RT-PCR
Prevalence and levels of Treponema denticola | baseline - 12 months
  Prevalence and levels of Treponema denticola, determined by means of RT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Claudio M Pannuti, PhD, Principal Investigator — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guglielmetti MR, Rosa EF, Lourencao DS, Inoue G, Gomes EF, De Micheli G, Mendes FM, Hirata RD, Hirata MH, Pannuti CM. Detection and quantification of periodontal pathogens in smokers and never-smokers with chronic periodontitis by real-time polymerase chain reaction. J Periodontol. 2014 Oct;85(10):1450-7. doi: 10.1902/jop.2014.140048. Epub 2014 May 2. PMID 24794687